CLINICAL TRIAL: NCT05882201
Title: Comparison of Femoral Nerve Block Versus Fascia Iliaca Compartment Block for Pain Control in Traumatic Femur Fracture Repair in Pediatric Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Mahdy Mohamed Elghanam, Principle investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2/2023ANESTH58
Record Dates: First submitted 2023-04-04; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Regional Anesthesia Morbidity

STUDY DESIGN:
Intervention Model Description: * The study will be a prospective randomized controlled study. Patients will be randomized by a computer-generated program into 3 equal parallel groups that will be randomly assigned to either:
  * Control group;(30 patient).
  * Group FICB; (30 patients) Fascia Iliaca compartment block group.
  * Group FNB; (30 patients) Femoral nerve block group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): Control group
  Interventions: Procedure: General care
- Group FICB (Experimental): ✓ Group FICB; (30 patients) Fascia Iliaca compartment block group.
  Interventions: Procedure: Fascia Iliaca compartment block group
- Group FNB (Experimental): ✓ Group FNB; (30 patients) Femoral nerve block group.
  Interventions: Procedure: Femoral nerve block group

INTERVENTIONS:
Procedure: Fascia Iliaca compartment block group — Group FICB Fascia: with the patient supine, the skin was prepped and draped with alcohol solution 70%,
  . A 22-G needle will be visualized entering the fascia Lata and the FI. bupivacaine, up to 2.5mg/kg of lean body weight with a volume of injectate of .5 ml/kg up to 40 ml will be injected after aspiration beneath the fascia Lata.
  Arms: Group FICB
Procedure: Femoral nerve block group — ✓ Group FNB; With the patient supine, the skin will be prepped and draped with alcohol solution 70% The nerve in the crosssection is a triangular white structure lateral to the femoral artery. Ultrasoundallows direct visualization of the needle and nerve as well as real-time monitoring of the injection of local anesthetic. An in-plane approach will be used to direct needle placement to the femoral nerve and inject after aspiration with bupivacaine, up to 2.5mg/kg of lean body weight with a volume of injectate of .5 ml/kg up to 40ml.
  Arms: Group FNB
Procedure: General care — using ordinary technique
  Arms: Control group

SUMMARY:
Pediatric orthopedic surgical procedures require a multimodal approach for anesthetic management that maximizes both patient comfort and safety.

(1) A multimodal strategy for perioperative pain management is often required for children undergoing orthopedic surgery including pharmacological methods, and regional anesthesia (R.A). (1,2) Recent guidelines published jointly by the European Society of Regional Anesthesia (ESRA) and the American Society of Regional Anesthesia (ASRA) recommend that regional blocks can and should preferably be performed under general anesthesia or deep sedation in children of all ages. (3,4) Many studies investigated the safety of regional pediatric nerve blocks These studies showed pediatric complication rates consistent with adult data. These complications include nerve injury, intravascular injection and local anesthetics systemic toxicity (LAST), and acute compartmental syndrome. these complications have been minimized by ultrasound-guided nerve block in pediatrics. (5) The annual incidence of pediatric femoral fractures is estimated to be 19 per 100,000. Femoral fractures are usually associated with other injuries such as intracranial hemorrhages, lung contusions, hemothorax or pneumothorax, and other organ injuries which make regional anesthesia (R.A) is preferable as a sole technique or combined with general anesthesia to decrease the overall dosage of anesthetics and opioids. (6) The most tangible advantage of RA is profound and prolonged pain relief. Alternatively, pain relief can be given by opioids which are known to cause nausea, vomiting, respiratory depression, decrease in gut motility and increase apneic spells in the population vulnerable to the same. Nonsteroidal anti- inflammatory drugs can affect the immature renal system adversely. RA offers pain relief without changing the physiological milieu. (7) Fascia iliaca Compartment Block (FICB) has been widely used for postoperative analgesia in patients undergoing hip, femoral bone, and knee surgical procedures. FICB was first introduced by Dalens et al in 1989. This regional plane block technique was used to block the femoral nerve and the lateral femoral cutaneous nerve of the thigh and the obturator nerve with a high level of safety and success, well-suited for the anterolateral surgeries of the thigh. (8,9) Femoral nerve block (FNB) has been widely used for postoperative analgesia in patients undergoing hip, and femoral bone surgical procedures, it provides anesthesia and analgesia for the lateral aspect of the thigh and the femur bone.

(10,11) FICB has a wider range of anesthesia and analgesia in lower limbs compared to FNB. but the use of dilute injectate in FICB may minimize sensory and motor block than FNB. (1,16) This study will be conducted to evaluate the effects of FICB vs FNB in pain control in pediatrics undergoing femoral fracture repair surgery.

DETAILED DESCRIPTION:
Pediatric orthopedic surgical procedures require a multimodal approach for anesthetic management that maximizes both patient comfort and safety.

(1) A multimodal strategy for perioperative pain management is often required for children undergoing orthopedic surgery including pharmacological methods, and regional anesthesia (R.A). (1,2) Recent guidelines published jointly by the European Society of Regional Anesthesia (ESRA) and the American Society of Regional Anesthesia (ASRA) recommend that regional blocks can and should preferably be performed under general anesthesia or deep sedation in children of all ages. (3,4) Many studies investigated the safety of regional pediatric nerve blocks These studies showed pediatric complication rates consistent with adult data. These complications include nerve injury, intravascular injection and local anesthetics systemic toxicity (LAST), and acute compartmental syndrome. these complications have been minimized by ultrasound-guided nerve block in pediatrics. (5) The annual incidence of pediatric femoral fractures is estimated to be 19 per 100,000. Femoral fractures are usually associated with other injuries such as intracranial hemorrhages, lung contusions, hemothorax or pneumothorax, and other organ injuries which make regional anesthesia (R.A) is preferable as a sole technique or combined with general anesthesia to decrease the overall dosage of anesthetics and opioids. (6) The most tangible advantage of RA is profound and prolonged pain relief. Alternatively, pain relief can be given by opioids which are known to cause nausea, vomiting, respiratory depression, decrease in gut motility and increase apneic spells in the population vulnerable to the same. Nonsteroidal anti- inflammatory drugs can affect the immature renal system adversely. RA offers pain relief without changing the physiological milieu. (7) Fascia iliaca Compartment Block (FICB) has been widely used for postoperative analgesia in patients undergoing hip, femoral bone, and knee surgical procedures. FICB was first introduced by Dalens et al in 1989. This regional plane block technique was used to block the femoral nerve and the lateral femoral cutaneous nerve of the thigh and the obturator nerve with a high level of safety and success, well-suited for the anterolateral surgeries of the thigh. (8,9) Femoral nerve block (FNB) has been widely used for postoperative analgesia in patients undergoing hip, and femoral bone surgical procedures, it provides anesthesia and analgesia for the lateral aspect of the thigh and the femur bone.

(10,11) FICB has a wider range of anesthesia and analgesia in lower limbs compared to FNB. but the use of dilute injectate in FICB may minimize sensory and motor block than FNB. (1,16) This study will be conducted to evaluate the effects of FICB vs FNB in pain control in pediatrics undergoing femoral fracture repair surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients are within the age range of 5 to 12 years old.
* Isolated Traumatic fracture of the femur bone.
* ASA I or II physical status.
* Pts weighed ≥10 kg

Exclusion Criteria:

* Refusal of the patient's parents or legal guardians to give informed consent.

  * History of allergy to any of the study drugs.
  * Injury at the site of injection.
  * Vascular compromise an injured leg.
  * Bilateral femur fracture.
  * Recent trauma to the head, chest, or abdomen.
  * history of bleeding disorder, or anticoagulant therapy.
  * Preoperative intake of opioid or non-steroidal anti-inflammatory drugs within 24 h before surgery.
  * Neurological and/or psychological diseases.
  * Associated cardio-respiratory illness.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | expected within 6 months
  Assessing the Postoperative pain using The Face, Legs, Activity, Cry and Consolability (FLACC) scale.

SECONDARY OUTCOMES:
Postoperative need for analgesia | expected within 6 months
  Postoperative need for analgesia using The visual analog scale (VAS) to evaluate the pain

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia university hospitails, Shibīn al Kawm, Menoufya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Wu JP. Pediatric Anesthesia Concerns and Management for Orthopedic Procedures. Pediatr Clin North Am. 2020 Feb;67(1):71-84. doi: 10.1016/j.pcl.2019.09.006. PMID 31779838